CLINICAL TRIAL: NCT01068756
Title: Effect of Rifampin on the Pharmacokinetics of Dapagliflozin in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: MB102-074
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dapagliflozin/Rifampin (Other)
  Interventions: Drug: Dapagliflozin; Drug: Rifampin

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, 10 mg, 2 single oral 10 mg doses, 2 days
Drug: Rifampin — Capsules, Oral, 600 mg, Once daily on days 4 to 11, 8 days

SUMMARY:
The purpose of the study is to assess the effects of rifampin on the pharmacokinetics of dapagliflozin

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Body Mass Index (BMI) of 18 to 32 inclusive
* Women who are not of childbearing potential and men, ages 18 to 45

Exclusion Criteria:

* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, electrocardiogram (ECG) or clinical laboratory determinations
* Glucosuria
* Abnormal liver function tests

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
AUC (area under the concentration-time curve) Single dose pharmacokinetic parameter will be derived from plasma concentration versus time data | Days 1 to 3 and Days 9 to 11

SECONDARY OUTCOMES:
Cmax (maximum observed concentration) Single dose pharmacokinetic parameter will be derived from plasma concentration versus time data | Days 1 to 3 and Days 9 to 11
Tmax (time of maximum observed concentration) Single dose pharmacokinetic parameter will be derived from plasma concentration versus time data | Days 1 to 3 and Days 9 to 11

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Ppd Development, Austin, Texas, United States

REFERENCES:
- See also: MB102-074_redacted_CSR_synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3652&filename=MB102-074_redacted_CSR_synopsis.pdf